CLINICAL TRIAL: NCT03002558
Title: Long-term Cardiovascular Outcomes in Patients With Resistant Hypertension and Obstructive Sleep Apnea With or Without Treatment With Continuous Positive Airway Pressure.
Brief Title: Long-term Cardiovascular Outcomes in Patients With RH and OSA With or Without Treatment With CPAP
Acronym: SARAH
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); ResMed (Industry)
Responsible Party: Principal Investigator, Ferran Barbe, MD, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: SARAH-1
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
Keywords: Hypertension; Continuous Positive Airway Pressure; Obstructive Sleep Apnea; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * 2 tubes EDTA
  * 2 tubes with gel for serum
  * 1 tube for RNA extraction
  * 1 tube for urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- control (non-OSA): Patients without sleep apnoea
- OSA-treated: Patients with sleep apnoea who are treated (CPAP, surgery or MAD)
- OSA-non treated: Patients with sleep apnoea who are not treated

SUMMARY:
Objectives:

Main objective: To assess the impact of obstructive sleep apnea (OSA) and its treatment on cardiovascular outcomes (morbidity and mortality) in patients with resistant hypertension (RH).

Secondary objectives: i) to identify the subclinical organ damage profile at baseline and its association with OSA, and to identify if long term blood pressure control and number of antihypertensive drugs needed is different depending on OSA diagnosis and its treatment; ii) to identify epigenetic profiles and clinical, biological and polygraphic variables with a predictive value for cardiovascular outcomes in RH patients with OSA; iii) to validate the HIPARCO-SCORE tool in men in an independent cohort and elaborate a new tool to be used in women; and iv) to perform a cost-effectiveness analysis to evaluate the impact of OSA diagnosis and treatment in patients with RH.

Methodology: Prospective cohort study. 1,371 RH patients will be recruited. Ambulatory blood pressure monitoring (ABPM), socio-demographic, clinical, OSA-related, biochemical and subclinical organ damage variables and biological samples at baseline will be collected from all the subjects included. A sleep study will be performed in all the subjects at the study inclusion date. Subsequently, the OSA subjects will be managed as per local standard practice. Follow-up variables will be annually collected (including blood samples). On the basis of OSA and its treatment, three cohorts of RH subjects will be defined: control (non-OSA), OSA-treated and OSA nontreated.

DETAILED DESCRIPTION:
A minimum follow-up of 5 years has been established. During the follow-up, an annually programmed visit will be carried on to all patients, collecting variables from subjects' interview in the office.The baseline and follow-up variables will be collected using questionnaires.

The variables that will be collected are:

BP variables; Anthropometric variables; Compliance with CPAP in the case of CPAP-treated OSA patients; blood samples extraction; outcomes (heart disease, cerebrovascular disease, kidney disease, vascular disease). All the cardiovascular events will be independently evaluated by two doctors to establish a diagnostic. In case of discordance a third external doctor will assess the case. The date of each event will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of RH according to the following criteria, which include 2 clinical situations: (i) BP above control in ABPM (24-h BP > 130/80 mmHg),regardless of optimal dose treatment with 3 agents (one must be a diuretic). Other causes of inadequate control must be discarded (poor compliance, drugs). (ii) Controlled BP but treated with no less than 4 medications.
* Patients aged 18 to 75 years old.
* To sign informed consent for the participation in the study.

Exclusion Criteria:

* Secondary hypertension to endocrinology causes (pheochromocytoma, Conn disease, Cushing´s Syndrome, hyperparathyroidism), drug treatment (NSAID or cortisone, immunodepressants, EPO), renal artery stenosis, alcohol abuse, aortic coarctation and intracranial tumours.
* Any process, that limits life expectancy to less than one year.
* Previously diagnosed OSA with current active treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Resistant Hypertension
Sampling Method: Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation the impact of OSA and its treatment on cardiovascular outcomes | After 5 years of follow-up
  OSA diagnosis shall be established by PSG or PCR. It will be evaluated cardiovascular outcomes (CV death, non-fatal acute myocardial infarction, non-fatal stroke, hospital admission for heart failure and new hospitalization for unstable angina or Transitory Ischemic Attack) before and after of OSA diagnosis and treatment.

SECONDARY OUTCOMES:
Cardiovascular composite: CV death, non-fatal acute myocardial infarction, non-fatal stroke, hospital admission for heart failure and new hospitalization for unstable angina or Transitory Ischemic Attack. | After 5 years of follow-up
  It will be evaluated cardiovascular outcomes at the end of the study. These outcomes will be collected from subjects' interviews at each yearly follow-up visit in the office and from computed medical records.
Identify epigenetic biomarkers signatures with a predictive value of favourable cardiovascular outcome in patients with RH. | After 5 years of follow-up
  Using DNA and RNA samples, it will be performed different analysis at the end of the study, to see if there is any change in genes related to both diseases
Validation the HIPARCO - Score tool in an independent cohort, men with resistant hypertension, OSA and CPAP compliance (≥4h/night) | 2 years
  Analyse mRNA to validate de HIPARCO score
Creation of a predictive tool (like HIPARCO-Score) for women | 3 years
  Identify a plasma miRNA profile that predicts blood pressure response to CPAP treatment.
Cost- Effectiveness analyses between study groups and to compare the cost of health care utilization between two year before and after the starting of the study related to the study groups. | After 5 years of follow-up
  Only direct costs will be considered. Analysis will include an estimation of quality-adjusted life-years (QALYs) gained

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé, Principal Investigator — Spanish Respiratory Society (SEPAR)
Locations (1):
- Spanish Respiratory Society, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sapina-Beltran E, Benitez ID, Torres G, Fortuna-Gutierrez AM, Ponte Marquez P, Masa JF, Drager LF, Cabrini M, Felez M, Vazquez S, Abad J, Lee C, Garcia-Rio F, Casitas R, Mediano O, Romero Peralta S, Martinez D, Sanchez-de-la-Torre M, Barbe F, Dalmases M. Effect of CPAP treatment on BP in resistant hypertensive patients according to the BP dipping pattern and the presence of nocturnal hypertension. Hypertens Res. 2022 Mar;45(3):436-444. doi: 10.1038/s41440-021-00762-7. Epub 2021 Dec 24. PMID 34952953
- [Derived] Sapina-Beltran E, Torres G, Benitez I, Fortuna-Gutierrez AM, Marquez PP, Masa JF, Corral-Penafiel J, Drager LF, Cabrini M, Felez M, Vazquez S, Abad J, Lee CH, Aung AT, Garcia-Rio F, Casitas R, Sanchez-de-la-Torre M, Gaeta AM, Barbe F, Dalmases M. Prevalence, Characteristics, and Association of Obstructive Sleep Apnea with Blood Pressure Control in Patients with Resistant Hypertension. Ann Am Thorac Soc. 2019 Nov;16(11):1414-1421. doi: 10.1513/AnnalsATS.201901-053OC. PMID 31514508